CLINICAL TRIAL: NCT07127133
Title: A Gait and Path Tortuosity System for Monitoring Cognitive Decline in Individuals at Risk for Alzheimer's Disease and/or Alzheimer's Disease Related Dementias (AD/ADRD)
Brief Title: An Insole and Ankle Device for Monitoring Cognitive Decline in Individuals at Risk for Alzheimer's Disease and/or Alzheimer's Disease Related Dementias (AD/ADRD)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Innovative Design Labs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: A24-016; R44AG063679 (NIH)
Record Dates: First submitted 2025-07-11; First posted 2025-08-17 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Mild Cognitive Impairment (MCI); Dementia
MeSH Terms: conditions — Cognitive Dysfunction; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Individuals using the insole and ankle device (Experimental): Participants will use the wearable leg module and insole device for either several hours in a lab environment or 1 week within their home and the community. Data will be recorded by the device
  Interventions: Device: Insole and ankle device

INTERVENTIONS:
Device: Insole and ankle device — Device that is worn as a shoe insole and around the ankle which will measure gait parameters to detect cognitive decline

SUMMARY:
This study tests an innovative system and service for collecting objective, consistent, and in-community gait parameters suitable for use as AD/ADRD biomarkers. The system is designed to be affordable, scalable, and practical for longitudinal, unsupervised, in-community use by older adults, including those with dementia symptoms. This study will be performed in two parts and involves collecting gait data from participants using the leg module and insole device either (1) for several hours in a lab setting (in-lab testing) or (2) within their home and community for 1 week (in-community testing). Thirty people who are healthy, have mild cognitive impairment, or who have Alzheimer's disease or related dementia will be recruited to participate in the in-lab testing, in which they will perform walking tasks and cognitive testing for several hours within a lab environment. After completion of in-lab testing, 120 individuals who are healthy, have mild cognitive impairment, or who have Alzheimer's disease or related dementia will be recruited to participate in the in-community testing, in which they will wear the insole and ankle device within their community for 1-week for collection of gait data in real world settings.

ELIGIBILITY:
Inclusion Criteria:

* Age 55 or older
* Ability to ambulate without the use of an assistive device. For this study, we will assume participants are ambulatory if they can complete the functional outcome measures (i.e., TUG) without the use of an assistive device
* Ability to understand and provide informed consent, or has a legally authorized representative (LAR) to provide consent on their behalf
* Ability to don and doff the insole and leg module independently or have assistance for the duration of the study

Exclusion Criteria:

* Non-English Speaking
* Use of ankle-foot orthosis for ambulation that prevents use of the system
* Self-reported acute thrombophlebitis including deep vein thrombosis
* Untreated lymphedema or lesion of any kind, swelling, infection, inflamed area of skin or eruptions on or near product use (foot and ankle)
* Untreated fractures in the foot and ankle
* Any other significant medical condition that may affect participation or performance in the study, as determined by investigators

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
In Lab Testing Primary Outcome: Mean absolute error of gait speed from the Short Physical Performance Battery and Timed Up and Go | Day 1
  Mean Absolute Error (MAE) of the gait speed during the Short Physical Performance Battery (SPPB) and Timed Up and GO (TUG)
In-Community Testing Primary Outcome: balanced accuracy of model developed using gait data | One week
  Balanced accuracy of cognitive impairment classification. This is the mean between recall of the positive and negative classes.

CONTACTS AND LOCATIONS:
Locations (1):
- HealthPartners Neuroscience Center, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No